CLINICAL TRIAL: NCT03511144
Title: A Prospective Randomised Double Blind Single Centre Study Comparing Measured Resection and Ligament Balancing Implantation Techniques Using the Unity Knee™ Total Knee System
Brief Title: A Comparison of Two Surgical Techniques Using the Unity Knee™ Total Knee System
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study not initiated
Sponsor: Corin (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CSP2015-04
Record Dates: First submitted 2018-04-11; First posted 2018-04-27 (Actual); Last update posted 2018-11-21 (Actual); Status verified 2018-11

CONDITIONS: Osteoarthritis, Knee; Rheumatoid Arthritis; Post-Traumatic Osteoarthritis of Knee; Varus Deformity, Not Elsewhere Classified, Knee; Valgus Deformity, Not Elsewhere Classified, Knee; Flexion Deformity, Knee; Fracture of Distal End of Femur; Fracture of Upper End of Tibia
MeSH Terms: conditions — Osteoarthritis, Knee; Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Measured resection (Active Comparator): Total knee replacement using the Unity Knee™ implanted with the measured resection surgical technique
  Interventions: Device: Unity Knee™ TKR using measured resection
- Ligament balancing (Active Comparator): Total knee replacement using the Unity Knee™ implanted with the ligament balancing surgical technique
  Interventions: Device: Unity Knee™ TKR using ligament balancing

INTERVENTIONS:
Device: Unity Knee™ TKR using measured resection — Total knee replacement using the Unity Knee™ implanted with the measured resection surgical technique
  Arms: Measured resection
Device: Unity Knee™ TKR using ligament balancing — Total knee replacement using the Unity Knee™ implanted with the ligament balancing surgical technique
  Arms: Ligament balancing

SUMMARY:
A comparison of two Unity Knee™ tissue-balancing techniques by analysing the results from X-rays and patient questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Subjects suitable for the Unity Knee™ Total Knee System according to the product "Instructions for use"
* Over 18 years old
* Male and female subjects who are skeletally mature
* Subjects who have a smartphone (iOS or Android) with internet connection via mobile Internet data or Wi-Fi connection
* Subjects able to understand what is expected of them and be able to comply with the study protocol requirements

Exclusion Criteria:

* Any subject listed for a revision total knee replacement or conversion of a unicondylar replacement to a total knee replacement on the operative knee
* Any subject with fixed flexion contracture greater than 20 degrees
* Any subject with varus/valgus deformity greater than 15 degrees
* Any subject with confirmed osteoarthritis or other pathologies affecting the contralateral knee that is anticipated to require surgery within 12 months
* Any subjects with contralateral knee replacement that is anticipated to require revision surgery within 12 months
* Any subject whose prospects for a recovery to independent mobility would be compromised by known co-existent, medical problems
* Any subject with a known sensitivity to device material
* Any subject who is pregnant
* Any subject currently a prisoner
* Any subject known to be a drug or alcohol abuser, or have a psychological disorder that could affect follow-up care or treatment outcomes
* Any subject currently involved in any personal injury litigation, medical-legal or worker's compensations claims
* Any subject unable to read and understand English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-07 (Estimated); Primary Completion 2019-09 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Posterior condylar offset (PCO) | 6 weeks post-op
  Any difference in PCO from preoperative to 6 weeks post-surgery

SECONDARY OUTCOMES:
Joint line in extension | 6 weeks post-op
  Any difference in vertical distance from medial epicondyle to distal medial femoral condyle articular surface from preoperative to 6 weeks post-surgery
Joint line in flexion | 6 weeks post-op
  Any difference in medial joint line position measured using the PCO
Femoral flexion angle | 6 weeks post-op
Distal femoral component angle | 6 weeks post-op
Tibial component angle | 6 weeks post-op
Tibial slope | 6 weeks post-op
Hip-knee-ankle (HKA) angle | 6 weeks post-op
Oxford Knee Score (OKS) | Up to 24 months post-op
Knee injury and Osteoarthritis Score - Physical Function Shortform (KOOS-PS) | Up to 24 months post-op
EuroQoL 5-dimension health state (EQ-5D 5-level) | Up to 6 months post-op
Hospital Anxiety and Depression Scale (HADS) | Up to 6 months post-op